CLINICAL TRIAL: NCT03877120
Title: Treatment Of Alcohol Withdrawal Syndrome: Dexmedetomidine Vs Diazepam In A Hospital O'horán
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centro Medico Nacional La Raza, IMSS (Other)
Collaborators: Universidad de La Frontera (Other)
Responsible Party: Principal Investigator, GARCIA MENDEZ NAYELY, Post doc Medical Sciences, Visiting professor, Universidad de la Frontera., Centro Medico Nacional La Raza, IMSS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEI-011-1-17
Record Dates: First submitted 2019-03-12; First posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Alcohol Withdrawal Delirium
Keywords: Dexmedetomidine; Diazepam; Alcohol dependence; Alcohol withdrawal syndrome; Benzodiacepines
MeSH Terms: conditions — Alcohol Withdrawal Delirium; Alcoholism | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Clinical Trials To compare Diazepam 5-20 mg IV or Dexmedetomidine 0.2-0.7 mcg / Kg / min., In monotherapy until the CIWA-Ar decreases to <10.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Sham Comparator): Dexmedetomidine. Dexmedetomidine use 400 mcg in 100 cc 0.9% physiological solution in continuous infusion starting at a dose of 0.2 mcg / kg / hr titrating until reaching a decrease in the adrenergic response, with a maximum dose of 0.7 mcg / kg / hr7.
  Dosage form: DEX 0.2-0.7 mcg/Kg/min.
  Interventions: Drug: Dexmedetomidine 0.004 MG/ML
- Diazepam (Active Comparator): Dosage form: Diazepam 5-10 mg IV, steps until a maximum dose of 120 mg diazepam
  Interventions: Drug: Diazepam Injectable Solution

INTERVENTIONS:
Drug: Dexmedetomidine 0.004 MG/ML — Experimental studies and single case reports suggest the α2-agonist dexmedetomidine is effective in managing the autonomic symptoms seen with alcohol withdrawal.
  Arms: Dexmedetomidine
Drug: Diazepam Injectable Solution — diazepam start with 5-20 mg IV as a dose response, steps until a maximum dose of 120 mg diazepam.
  Arms: Diazepam

SUMMARY:
The cessation of alcohol consumption of people suffering from alcohol abuse frequently leads to the development of an alcohol withdrawal syndrome (AWS).

The ethylic suppression syndrome is defined as the appearance of two or more data of autonomic hyperactivity, nausea, hallucinations and seizures associated with the cessation of alcohol consumption. For its evaluation, the CIWA-Ar scale is used, which guides the treatment based on benzodiazepines but with many adverse effects, so sedatives have been tried, among them dexmedetomidine, an alpha-agonist with action in the locus caeruleus, with variable results. Objectives: The investigators aimed to compare the DEX vs. Diazepam, for moderate disease, applying the CIWA-Ar scale, in participants with severe to moderate AWS. Methodology: 40 participants with CIWA-Ar greater than 10 points, the investigators are collected and randomized into two groups: one under treatment with diazepam (Group Diazepam) and another with dexmedetomidine (Group Dexmedetomidine), until the CIWA-Ar was reduced to less than 10, and adverse effects the investigators also reported. The analysis was done with student t. Results: The average duration of treatment with diazepam was 5.5 days (IC 95 = 6.6-3.8), the average duration of treatment with dexmedetomidine was 3.1 days (95% CI = 4.5-1.7), with a significant difference ( p = 0.0016). In the group with diazepam 60% presented adverse effects and in the group with dexmedetomidine 25% presented them, with a significant difference (p = 0.04). Conclusion: dexmedetomidine was superior to diazepam for the treatment of moderate-severe alcohol withdrawal with fewer adverse effects.

KEY WORDS: Alcohol dependence · Alcohol withdrawal syndrome · Dexmedetomidine · Diazepam · Benzodiazepines

DETAILED DESCRIPTION:
Alcohol withdrawal syndrome AWS (Alcohol Withdrawal Syndrome), is defined as the appearance of two or more data of autonomic hyperactivity, nausea, hallucinations and seizures associated with cessation of alcohol consumption. For its evaluation, the CIWA-Ar (Clinical Institute Withdrawal Assessment for Alcohol) scale is used, which guides the treatment based on benzodiazepines but a disadvantage is the related adverse effects, for which other pharmacological strategies of sedation have been tried, among them Dexmedetomidine (DEX).

OBJECTIVES:

The investigators aimed to compare the DEX vs. Diazepam, for moderate disease, applying the CIWA-Ar scale, in participants with severe to moderate AWS (Alcohol Withdrawal Syndrome).

MATERIALS:

Prior authorization from the ethics committee of O'Horán Hospital, Yucatán, Mexico. No. Registration CEI-011-1-17, and signature of informed consent. A randomized clinical trial was carried out in the Adult Emergencies service during the period July 2017-July 2018. Forty participants with CIWA-Ar greater than 10 points participated. The administration of:

A) Diazepam 5-20 mg IV. B) DEX 0.2-0.7 mcg / Kg / min., until the CIWA-Ar scale decreases to <10.

The investigators are excluded minor patients, mild CIWA-Ar category, previous medication, participants with severe cranial encephalic trauma (TBI) or mechanical ventilation requirement, with chronic liver failure category C in the Child-Turcotte-Pugh classification.

RESULTS

The CIWA Ar scale average for admission was 23 points, the lowest of 10 points and the highest of 38 points. The average number of days consuming alcohol prior to hospital admission was 131.9, with the highest average in the group that used dexmedetomidine; the average number of days after having suspended the intake until hospital admission was 1.7 days, being slightly higher in the group that used diazepam; the shortest time was 6 hours and the longest of a week without being related to the CIWA Ar score.

The average duration of treatment with diazepam was 5.5 days (IC 95 = 6.6-3.8), The average duration of treatment with dexmedetomidine was 3.1 days (95% CI = 4.5-1.7) After applying t student a significant difference was found in the number of days in favor of dexmedetomidine (p = 0.0016)

CONCLUSIONS

The investigators found that DEX at conventional doses, for the treatment of moderate-severe alcohol withdrawal in terms of reducing the CIWA-Ar scale, in fewer days and with fewer adverse effects and complications.

REFERENCES:

1. Anderson P, Lars M, Gauden G. Alchol in the Europen Union. Consume, harm and policy approaches. Edit. WHO. 2012
2. Nota descriptiva N° 349: Alcohol. Organización Mundial de la Salud. 2015.
3. Encuesta Nacional de Adicciones 2011: Reporte de Alcohol. Medina-Mora ME, Villatoro-Velázquez JA, Fleiz-Bautista C, et. Al. México: INPRFM; 2012.
4. Longo D, Fauci A, Kasper E, et al. Harrison: Principios de Medicina Interna. 18ª ed. McGraw-Hill. México. 2012.
5. Diagnostic and statistical manual of mental disorders. 5th edition. Washington, DC: American Psychiatric Association; 2013. 947 pp.
6. Carson L, Kumar N, Wong-Mckinstry. Alcohol Withdrawal Syndrome. Critical Care. 2012.
7. Jawa R, Stothert J, Shostrom V, et al. Alcohol Withdrawal Syndrome in admitted trauma patients. The American Journal of Surgery (2014)208: 781-787
8. Sullivan J, Sykora K, Schneiderman J, et al. Assessment of alcohol withdrawal: the revised clinical institute withdrawal assessment for alcohol scale (CIWA-Ar). Br J Addict. 1989. 84(11):1353-7.
9. Waye C, Wong M, Lee S. Implementation of a CIWA Ar Alcohol Withdrawal protocol in a Veterans Hospital. South Med Jour. 2015. 108(1):23-8.
10. Ramírez D, Sánchez G. Capacidad diagnóstica de las escalas de Cushman y AWS para supresión etílica. Med Int de Mex. 2013. 29(1): 26-31
11. Miller W, McCurdy L. A double-blind comparison of the efficacy and safety of lorazepam and diazepam in the treatment of the acute alcohol withdrawal syndrome. Clin Ther 1984. 6(3):364-71.
12. Henrey G, Dery R, Bandes R. A prospective randomized trial of phenobarbital vs benzodiazepines for acute alcohol withdrawal. Am Jour Eme Med. 2011. 382-85.
13. Hughes D, VanWert E, LePori L. Propofol for benzodiazepine-refractory alcohol withdrawal in a non-mechanically ventilated patient. Am Jour Eme Med. 2014. 112.e3-e4.
14. Wong A, et al. Multicenter evaluation of pharmacologic management and outcomes associated with severe resistant alcohol withdrawal. J Crit Care. 2014.
15. Samuels E, Szabadi E. Functional Neuroanatomy of the Noradrenergic Locus Coeruleus: Its Roles in the Regulation of Arousal and Autonomic Function Part I: Principles of Functional Organisation. Curr Neuropharmacol. 2008; 6(3): 235-53.
16. Rovasalo A, Tohmo H, Aantaa R, Kettunen E, Palojoki R: Dexmedetomidine as an adjuvant in the treatment of alcohol withdrawal delirium: a case report. Gen Hosp Psychiatr 2006, 28:362-363.
17. Rayner et al. Dexmedetomidine as adjunct treatment for severe alcohol withdrawal. Annasl of intensive care. 2012. 2:12
18. VanderWeid L, Foster C, McLaren R. Evaluation of early dexmedetomidine addition to the standard of care for severe alcohol withdrawal in the ICU: A retrospective controlled cohort study. Jour Int Care Med. 2014. 1-7.
19. Frazee E, Personett H, Leung J, et al. Influence of dexmedetomidine therapy on the management of severe alcohol withdrawal síndrome in critically ill patients. Jour Crit Care. 2014. 198-302.
20. Crispo A, Daley M, Pepin J. Comparison of clinical outcomes in nonintubated patients with severe alcohol withdrawal síndrome treated with continuous-infusion sedatives: dexmedetomidine versus benzodiazepines. Pharm. 2014. 910-17.
21. Pita S. Determinación del tamaño muestreal. Cad Aten Prim. 1996. 138-44.
22. Farmacología Básica y clínica. P Lorenzo, A Moreno, Lizasoain, et al. 18ª ed. Editorial Panamericana. España. 2010.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received dexmedetomidine during their Emergency stay
* Patients who received diazepam during their Emergency stay
* CIE-10 codes consistent with alcohol withdrawal during hospitalization
* CIWA-A score >10 points

Exclusion Criteria:

* comorbid disease, including several with CNS trauma or cerebrovascular accidents, one with end-stage metastatic carcinoma, and one patient with severe sepsis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 2 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Average Alcohol Withdrawal Scoring | dosing, total dose per 24 hours period for each patient, limited to 10 days
  Total Score = 0 - 9: absent or minimal withdrawal 10 - 19: mild to moderate withdrawal more than 20: severe withdrawal
Average Diazepam Received (mg) | Limited to 10 days
  Dosis total: Diacepam 5-20 mg IV
Average Dexmedetomidine Received (mg) | dosing, total dose per 24 hours period for each patient, limited to 10 days
  Infusión: DEX 0.2-0.7 mcg/Kg/min
heart rate average | 24 hours
  mean values per 24 hours period for each patient
Systolic blood pressure average | 24hours
  mean values per 24 hours period for each patient

SECONDARY OUTCOMES:
days of hospital stay | 24 hours limited to 10 days
  Duration in days of hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Nayely Garcia Mendez, Mexico City, Mexico

REFERENCES:
- [Result] Yost DA. Alcohol withdrawal syndrome. Am Fam Physician. 1996 Aug;54(2):657-64, 669. PMID 8701843
- [Derived] Garcia-Mendez N, Briceno-Santana M, Totomoch-Serra A, Manterola C, Otzen T, Valdez PS, Campos-Duran R, Reyna GC. The hemodynamic effects of diazepam versus dexmedetomidine in the treatment of alcohol withdrawal syndrome: A randomized clinical trial. Med Clin (Barc). 2021 Dec 24;157(12):561-568. doi: 10.1016/j.medcli.2020.09.023. Epub 2021 Jan 8. English, Spanish. PMID 33423824